CLINICAL TRIAL: NCT04181190
Title: Effects of Anti-IL5 Biological Treatments of Total Blood IgE Levels in Severe Asthmatic Patients: Real-life Retrospective Multicenter Observational Study
Brief Title: Effects of Anti-IL5 Biological Treatments on Blood IgE Levels in Severe Asthmatic Patients
Acronym: BIONIGE
Status: Completed | Type: Observational
Sponsor: Università degli Studi di Ferrara (Other)
Responsible Party: Principal Investigator, Alberto Papi, MD, Head of Respiratory Unit, Università degli Studi di Ferrara
Other Study IDs: 272/2019/Oss/AOUFe BIONIGE
Record Dates: First submitted 2019-11-15; First posted 2019-11-29 (Actual); Last update posted 2020-11-04 (Actual); Status verified 2020-11

CONDITIONS: Asthma; Asthma; Eosinophilic
Keywords: IgE; Eosinophils; Mepolizumab; Benralizumab; Severe Asthma
MeSH Terms: conditions — Asthma; Pulmonary Eosinophilia | interventions — Blood Cell Count; Respiratory Function Tests

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Mepolizumab group: atopic patients with severe eosinophilic asthma treated with anti-IL-5 monoclonal antibody (Mepolizumab)
  Interventions: Diagnostic Test: Total IgE; Diagnostic Test: Blood cell counts; Diagnostic Test: Asthma control assessment; Diagnostic Test: lung function tests
- Benralizumab group: atopic patients with severe eosinophilic asthma treated with anti-IL5 receptor monoclonal antibody (Benralizumab)
  Interventions: Diagnostic Test: Total IgE; Diagnostic Test: Blood cell counts; Diagnostic Test: Asthma control assessment; Diagnostic Test: lung function tests

INTERVENTIONS:
Diagnostic Test: Total IgE — Levels of total IgE before biological treatments and at 4±2 months of treatments
Diagnostic Test: Blood cell counts — White Blood Cell Count and Differential (and in particular the levels of total leucocytes, lymphocytes, eosinophils and basophils)
Diagnostic Test: Asthma control assessment — Levels of asthma control assessed by asthma control questionnaire (ACT) before initiation of biological treatments and at 4± months of treatments
Diagnostic Test: lung function tests — Lung function tests performed before initiation of biological treatments and at 4± months of treatments

SUMMARY:
Real-life, observational, retrospective, multicenter study to evaluate the effects of anti-IL5 biological treatments on blood total IgE Levels in atopic patients with severe eosinophilic asthma.

DETAILED DESCRIPTION:
Severe asthma, i.e. asthma that is not controlled despite maximal optimized therapy and/or that worsens when high dose treatment is decreased (GINA guidelines - available at https://ginasthma.or), is a major unmet medical need. Major advances in the management of severe asthma occurred in the past few years due to the new targeted biological therapies. Mepolizumab and Benralizumab are humanized monoclonal antibodies able to block interleukin (IL)-5 and the receptor for IL-5, respectively. These biological treatments block the eosinophilic driven inflammation. The effects of these treatments on an other key effector molecule of the T2-immune response, i.e. IgE, is virtually unknown.

To explore this issue, we set up a real life, observational, retrospective, multicenter study. The study will enroll patients with severe eosinophilic asthma already treated with Mepolizumab or Benralizumab. The following variable will be collected before the the biological treatment and at 4±2 months after the initiation of the pharmacological regimen:

* demographic data
* age of onset of asthma
* smoking habit
* concomitant pharmacological regimens
* number of asthma exacerbations since last visit
* concomitant diseases (particularly gastroesophageal reflux, nasal polyposis, atopic dermatitis, obesity, anxiety-depressive syndrome).
* White Blood Cell Count and Differential (and in particular the levels of total leucocytes, lymphocytes, eosinophils and basophils)
* Lung function tests (spirometry)

ELIGIBILITY:
Inclusion Criteria:

* atopy
* severe eosinophilic asthma (according to GINA guideline - available at https://ginasthma.org)
* patients treated with monoclonal antibody anti IL-5 (Mepolizumab) or with IL-5 anti-receptor monoclonal antibody (Benralizumab).
* stable asthma (free from asthma exacerbation for at least 8 weeks)

Exclusion Criteria:

* asthma exacerbation in last 8 weeks
* patients treated for COPD

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: atopic patients with severe eosinophilic asthma treated with anti IL-5 (Mepolizumab) or anti IL5-receptor (Benralizumab) humanized monoclonal antibodies
Sampling Method: Non-Probability Sample
Enrollment: 130 (Actual)
Dates: Start 2019-10-11 (Actual); Primary Completion 2020-10-01 (Actual); Study Completion 2020-11-01 (Actual)

PRIMARY OUTCOMES:
IgE levels in mepolizumab group | 4±2 months
  To evaluate total IgE levels (kU/l) in atopic patients with severe eosinophilic asthma at baseline and at 4 ± 2 months after initiation of anti-IL5 monoclonal antibody Mepolizumab

SECONDARY OUTCOMES:
Total leucocytes in mepolizumab group | 4±2 months
  To evaluate total leucocytes (number of cell/µl) in atopic patients with severe eosinophilic asthma at baseline and at 4 ± 2 months from the start of treatment with anti-IL5 monoclonal antibody Mepolizumab
Eosinophils (number) in mepolizumab group | 4±2 months
  To evaluate the number of blood eosinophils (cell/µl) in atopic patients with severe eosinophilic asthma at baseline and at 4 ± 2 months from the start of treatment with anti-IL5 monoclonal antibody Mepolizumab
Eosinophils (%) in mepolizumab group | 4±2 months
  To evaluate the percentage of blood eosinophils (%) total blood white cells in atopic patients with severe eosinophilic asthma at baseline and at 4 ± 2 months from the start of treatment with anti-IL5 monoclonal antibody Mepolizumab
Basophils (number) in mepolizumab group | 4±2 months
  To evaluate the number of blood basophils (cell/µl) in atopic patients with severe eosinophilic asthma at baseline and at 4 ± 2 months from the start of treatment with anti-IL5 monoclonal antibody Mepolizumab
Basophils (%) in mepolizumab group | 4±2 months
  To evaluate the percentage of blood basophils (%) to totale white blood cells in atopic patients with severe eosinophilic asthma at baseline and at 4 ± 2 months from the start of treatment with anti-IL5 monoclonal antibody Mepolizumab
lymphocytes (number) in mepolizumab group | 4±2 months
  To evaluate the number of blood lymphocytes (cell/µl) in atopic patients with severe eosinophilic asthma at baseline and at 4 ± 2 months from the start of treatment with anti-IL5 monoclonal antibody Mepolizumab
Lymphocytes (%) in mepolizumab group | 4±2 months
  To evaluate the percentage of blood lymphocytes (%) to total white cells in atopic patients with severe eosinophilic asthma at 4 ± 2 months from the start of treatment with anti-IL5 monoclonal antibody Mepolizumab
IgE levels in Benralizumab group | 4±2 months
  To evaluate total IgE levels (kU/l) in atopic patients with severe eosinophilic asthma at baseline and at 4 ± 2 months from the start of treatment with Benralizumab
Total leucocytes in Benralizumab group | 4±2 months
  To evaluate total leucocytes (number of cell/µl) in atopic patients with severe eosinophilic asthma at baseline and at 4 ± 2 months from the start of treatment with Benralizumab compared to the pretreatment value
Eosinophils (number) in Benralizumab group | 4±2 months
  To evaluate the number of blood eosinophils (cell/µl) in atopic patients with severe eosinophilic asthma at baseline and at 4 ± 2 months from the start of treatment with Benralizumab
Eosinophils (%) in Benralizumab group | 4±2 months
  To evaluate the percentage of blood eosinophils (%) total blood white cells in atopic patients with severe eosinophilic asthma at baseline and at 4 ± 2 months from the start of treatment with Benralizumab
Basophils (number) in Benralizumab group | 4±2 months
  To evaluate the number of blood basophils (cell/µl) in atopic patients with severe eosinophilic asthma at baseline and at 4 ± 2 months from the start of treatment with Benralizumab
Basophils (%) in Benralizumab group | 4±2 months
  To evaluate the percentage of blood basophils (%) to totale white blood cells in atopic patients with severe eosinophilic asthma at baseline and at 4 ± 2 months from the start of treatment with Benralizumab
Lymphocytes (number) in Benralizumab group | 4±2 months
  To evaluate the number of blood lymphocytes (cell/µl) in atopic patients with severe eosinophilic asthma at baseline and at 4 ± 2 months from the start of treatment with Benralizumab
Lymphocites (%) in Benralizumab group | 4±2 months
  To evaluate the percentage of blood lymphocytes (%) to total white cells in atopic patients with severe eosinophilic asthma at 4 ± 2 months from the start of treatment with Benralizumab
respiratory function (FEV1 - liter) in Mepolizumab group | 4±2 months
  To evaluate FEV1 (liter) in patients with severe eosinophilic asthma at baseline and at 4 ± 2 months from the start of treatment with Mepolizumab
respiratory function (FEV1 - %) in Mepolizumab group | 4±2 months
  To evaluate FEV1 (% predicted) in patients with severe eosinophilic asthma at baseline and at 4 ± 2 months from the start of treatment with Mepolizumab
respiratory function (vital capacity - liter) in Mepolizumab group | 4±2 months
  To evaluate vital capacity (VC - liter) in patients with severe eosinophilic asthma at baseline and at 4 ± 2 months from the start of treatment with Mepolizumab
respiratory function (vital capacity - %) in Mepolizumab group | 4±2 months
  To evaluate VC (% predicted) in patients with severe eosinophilic asthma at baseline and at 4 ± 2 months from the start of treatment with Mepolizumab
respiratory function (forced vital capacity - liter) in Mepolizumab group | 4±2 months
  To evaluate forced vital capacity (FVC - liter) in patients with severe eosinophilic asthma at baseline and at 4 ± 2 months from the start of treatment with Mepolizumab
respiratory function (forced vital capacity - % predicted) in Mepolizumab group | 4±2 months
  To evaluate FVC (% predicted) in patients with severe eosinophilic asthma at baseline and at 4 ± 2 months from the start of treatment with Mepolizumab
respiratory function (FEV1/FVC ratio) in Mepolizumab group | 4±2 months
  To evaluate FEV1/FVC ratio in patients with severe eosinophilic asthma at baseline and at 4 ± 2 months from the start of treatment with Mepolizumab compared to the pretreatment value.
respiratory function (FEV1/VC ratio) in Mepolizumab group | 4±2 months
  To evaluate FEV1/VC ratio in patients with severe eosinophilic asthma at baseline and at 4 ± 2 months from the start of treatment with Mepolizumab
respiratory function (FEV1 - %) in Benralizumab group | 4±2 months
  To evaluate FEV1 (% predicted) in patients with severe eosinophilic asthma at baseline and at 4 ± 2 months from the start of treatment with Benraluzumab
respiratory function (FEV1 - lier) in Benralizumab group | 4±2 months
  To evaluate FEV1 (liter) in patients with severe eosinophilic asthma at baseline and at 4 ± 2 months from the start of treatment with Benraluzumab
respiratory function (FVC - liter) in Benralizumab group | 4±2 months
  To evaluate FVC (liter) in patients with severe eosinophilic asthma at baseline and at 4 ± 2 months from the start of treatment with Benraluzumab
respiratory function (FVC - %) in Benralizumab group | 4±2 months
  To evaluate FVC (% predicted) in patients with severe eosinophilic asthma at baseline and at 4 ± 2 months from the start of treatment with Benraluzumab
respiratory function (VC - liter) in Benralizumab group | 4±2 months
  To evaluate VC (liter) in patients with severe eosinophilic asthma at baseline and at 4 ± 2 months from the start of treatment with Benraluzumab
respiratory function (VC - %) in Benralizumab group | 4±2 months
  To evaluate VC (% predicted) in patients with severe eosinophilic asthma at baseline and at 4 ± 2 months from the start of treatment with Benraluzumab
respiratory function (FEV1/FVC ratio) in Benralizumab group | 4±2 months
  To evaluate FEV1/VC ratio in patients with severe eosinophilic asthma at baseline and at 4 ± 2 months from the start of treatment with Benraluzumab compared to the pretreatment value.
respiratory function (FEV1/VC ratio) in Benralizumab group | 4±2 months
  To evaluate FEV1/FVC ratio in patients with severe eosinophilic asthma at baseline and at 4 ± 2 months from the start of treatment with Benraluzumab
Fractional exhaled nitric oxigen (FeNO) in Mepozumab group | 4±2 months
  To evaluate FeNO (ppb) in patients with severe eosinophilic asthma at baseline and at 4 ± 2 months from the start of treatment with Mepolizumab
Fractional exhaled nitric oxigen (FeNO) in Benralizumab group | 4±2 months
  To evaluate FeNO (ppb) in patients with severe eosinophilic asthma at baseline and at 4 ± 2 months from the start of treatment with Benraluzumab
Asthma control test in Mepolizumab group | 4±2 months
  To evaluate asthma control test (ACT) in patients with severe eosinophilic asthma at baseline and at baseline and at 4 ± 2 months from the start of Mepolizumab
Asthma control test in Benralizumab group | 4±2 months
  To evaluate asthma control test (ACT) in patients with severe eosinophilic asthma at baseline and at baseline and at 4 ± 2 months from the start of Benralizumab
correlation between eosinophils and total IgE | 4±2 months
  To evaluate the correlations (Pearson correlation coefficient) between the change in total eosinophil counts and IgE levels in patients treated with Mepolizumab or Benralizumab.
correlation between total IgE and lung function | 4±2 months
  To evaluate the correlations (Pearson correlation coefficient) between the change in total IgE levels and in functional parameters (FEV1, FVC and VC) in patients treated with Mepolizumab or Benralizumab.
correlation between total IgE and asthma control | 4±2 months
  To evaluate the correlations (Pearson correlation coefficient) between the change in total IgE levels and the change of asthma control (measured by asthma control test - ACT) in patients treated with Mepolizumab or Benralizumab.

CONTACTS AND LOCATIONS:
Overall Officials: Marco Contoli, Prof, Principal Investigator — Università di Ferrara - Azienda Ospedaliero Universitaria di Ferrara
Locations (8):
- Italy (8):
  - Azienda Ospedaliero Universitaria Ferrara, Ferrara
  - Professor of Respiratory Medicine Department of Medical and Surgical Sciences University of Foggia - Italy, Foggia
  - UOC Pneumologia Ospedale L.Sacco - Polo Univestiario ASST Fatebenefratelli - Milano, Milan
  - Malattie dell' Apparato Respiratorio Dipartimento di Scienza Mediche e Chirurgiche Materni-Infantili e dell'Adulto. Azienda Ospedaliero Universitaria di Modena, Modena
  - AOUP Giaccone Palermo, dipartimento PROMISE, Università di Palermo, Palermo
  - S.C di Pneumologia Ospedale S. Maria degli Angeli AAS5 Friuli Occidentale, Pordenone
  - Department of Medical Specialties, Pneumology Unit, Arcispedale Santa Maria Nuova, Azienda USL di Reggio Emilia-IRCCS, Reggio Emilia
  - UOC Pneumologia Azienda Ospedaliera Univeristaria Integrata - Verona, Verona

IPD SHARING:
Plan to Share IPD: Undecided